CLINICAL TRIAL: NCT03459105
Title: Ultrasound-assisted Versus Conventional Landmark-guided Spinal Anesthesia in Patients With Abnormal Spinal Anatomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1801-107-917
Record Dates: First submitted 2018-02-27; First posted 2018-03-08 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia, Spinal; Ultrasonography; Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Congresses as Topic; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-assisted (Experimental): Preprocedural ultrasound-assisted paramedian spinal anesthesia will be performed. 0.5% heavy bupivacaine will be injected to intrathecal space for spinal anesthesia.
  Interventions: Procedure: Ultrasound-assisted paramedian spinal anesthesia; Drug: 0.5% heavy bupivacaine
- Landmark-guided (Active Comparator): Landmark-guided spinal anesthesia will be performed, via either midline or paramedian approach. 0.5% heavy bupivacaine will be injected to intrathecal space for spinal anesthesia.
  Interventions: Procedure: Landmark-guided spinal anesthesia; Drug: 0.5% heavy bupivacaine

INTERVENTIONS:
Procedure: Ultrasound-assisted paramedian spinal anesthesia — A preprocedural ultrasound scanning will be done, and skin marking will be made. The needle entry point and insertion angle will be determined based on ultrasound scanning. Spinal anesthesia will be performed via paramedian approach.
  Other Names: sono-assisted
  Arms: Ultrasound-assisted
Procedure: Landmark-guided spinal anesthesia — Spinal anesthesia will be done using conventional landmark-guided technique.
  Other Names: conventional
  Arms: Landmark-guided
Drug: 0.5% heavy bupivacaine — 0.5% heavy bupivacaine will be administered into intrathecal space. The dose of local anesthetic injected for spinal anesthesia will be at the discretion of the attending anesthesiologist. The dose range of intrathecal bupivacaine will be between 12 and 16 mg.
  Other Names: bupivacaine

SUMMARY:
Spinal anesthesia can be challenging in patients with lumbar scoliosis or previous lumbar spine surgery. This study aims to evaluate whether the use of the ultrasound-assisted spinal anesthesia reduces the number of passes required to successful dural puncture compared with the conventional surface landmark-guided technique in patients with abnormal spinal anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergoing elective orthopedic surgery under spinal anesthesia,
* with ASA physical status classification I, II, III,
* and with (1) or (2)

  1. documented scoliosis in preoperative L-S-Spine X-ray (Cobb abgle > 10 degree)
  2. previous history of lumbar spinal surgery

Exclusion Criteria:

* Patients with contraindication to spinal anesthesia (coagulopathy, local infection, allergy to local anesthetic)
* Patients with morbid cardiac diseases
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
the number of needle passes | Intraoperative (from the first insertion of needle to patient's skin, until the completion of spinal anesthetic injection)
  the number of forward advancements of the spinal needle in a given interspinous space, i.e., withdrawal and redirection of spinal needle without exiting the skin

SECONDARY OUTCOMES:
Number of spinal needle insertion attempts | Intraoperative (from the first insertion of needle to patient's skin, until the completion of spinal anesthetic injection)
  the number of times the spinal needle was withdrawn from the skin and reinserted
Time for identifying landmarks | 1 day (time taken for establish the landmark, from start of palpation/US scanning to completion of palpation/scanning)
  In group L, time from start of palpation to completion of the process, as declared by the anesthesiologist. In group U, time from placement of the ultrasound probe on the skin to the completion of markings.
Time taken for performing spinal anesthetic | Intraoperative (from insertion of the needle to the completion of injection)
  time from needle insertion to the completion of injection
dermatome level of sensory block | 5, 10, 15 minutes after the completion of spinal anesthetic injection
  thoracic dermatome level of sensory block assessed by loss of cold sensation tested with 2% chlorhexidine swab
Incidence of radicular pain, paraesthesia, and blood tapping in the spinal needle | Intraoperative (from the first insertion of needle, until the completion of spinal anesthetic injection)
  Incidence of radicular pain, paraesthesia, and blood tapping in the spinal needle during the spinal anesthesia procedure
Periprocedural pain | Patients will be asked immediately after the completion of spinal anesthesia
  11-point verbal rating scale (0=no pain, 10=most pain imaginable)
Periprocedural discomfort score | Patients will be asked immediately after the completion of spinal anesthesia
  11-point verbal rating scale (0=no discomfort, 10=most discomfort imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316